CLINICAL TRIAL: NCT06249347
Title: Pulmonary Vein Isolation and Left Roof Linear, Mitral Isthmus Linear, and Left Anterior Septal Linear Ablation, and Left Atrial Appendage Device Occlusion in Patients With Non-paroxysmal Atrial Fibrillation: PROMISED Trial.
Brief Title: Left Roof Linear, Mitral Isthmus Linear and Left Anterior Septal Linear Ablation for Non-paroxysmal AF: PROMISED Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2024-01-104
Record Dates: First submitted 2024-01-08; First posted 2024-02-08 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation, Persistent
Keywords: non-paroxysmal atrial fibrillation; left atrial anterior wall ablation; roof linear ablation; mitral isthmus linear ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Cases were prospectively treated in a 2-arm 1:1 design according to ablation strategy, divided into the Promised group (n = 83) or the PVI combined LAAC group (n =83).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROMISED (Experimental): Guided by a circular mapping catheter, all patients initially underwent wide-area circumferential pulmonary vein isolation (CPVI) using radiofrequency ablation catheter. If sinus rhythm was restored after performing the CPVI ablation, the ablation procedure would be stopped. If AF persisted, patients underwent linear ablation (roof linear ablation+anterior septal linear ablation+mitral isthmus linear ablation) using radiofrequency ablation catheter. Then, guided by left atrial appendage (LAA) angiography, the operators selected an appropriately sized left atrial appendage occlusion device according to the LAA size and morphology.
  Interventions:
  Procedure: CPVI+ roof linear ablation + anterior septal linear ablation + mitral isthmus linear ablation + Left atrial appendage closure (LAAC)
  Interventions: Procedure: PROMISED; Device: Radiofrequency ablation catheter; Device: left atrial appendage occlusion device
- CPVI and LAAC (Active Comparator): Guided by a circular mapping catheter, all patients initially underwent wide-area CPVI using radiofrequency ablation catheter. Then, guided by LAA angiography, the operators selected an appropriately sized left atrial appendage occlusion device according to the LAA size and morphology.
  Interventions:
  Procedure: CPVI and LAAC
  Interventions: Procedure: CPVI and LAAC; Device: Radiofrequency ablation catheter; Device: left atrial appendage occlusion device

INTERVENTIONS:
Procedure: PROMISED — CPVI: Achievement of a wide disconnection of the right and left pulmonary veins; Roof linear ablation: linear ablation in the left atria roof; Anterior septal linear ablation: linear ablation in the anterior septal linear which coursed from the middle of the right superior and inferior pulmonary veins or the middle of the right superior pulmonary vein to the mitral valve annulus; Mitral isthmus linear ablation: linear ablation in the mitral isthmus; Left atrial appendage closure: Occlusion of the left atrial appendage with a left atrial appendage occlusion device.
  Arms: PROMISED
Procedure: CPVI and LAAC — CPVI: Achievement of a wide disconnection of the right and left pulmonary veins; Left atrial appendage closure: Occlusion of the left atrial appendage with a left atrial appendage occlusion device.
  Arms: CPVI and LAAC
Device: Radiofrequency ablation catheter — Device： Radiofrequency ablation catheter
Device: left atrial appendage occlusion device — Device： left atrial appendage occlusion device

SUMMARY:
The purpose of this prospective randomized study is to assess whether a new treatment strategy consisting of circumferential Pulmonary vein isolation (PVI), left ROof linear (RL), Mitral Isthmus linear (MIL), and left anterior SEptal linear (ASL) ablation and left atrial appendage (LAA) Device occlusion (PROMISED procedure) is superior to the PVI combined LAA closure in enhancing the long-term success rate of catheter ablation in non-paroxysmal atrial fibrillation (AF) patients.

DETAILED DESCRIPTION:
Circumferential pulmonary vein isolation (CPVI) is an important radiofrequency catheter ablation strategy for AF. The recurrence rate of non-paroxysmal AF (non-PAF) after CPVI remains unsatisfactory, despite the use of additional strategies, such as linear ablation and complex fractionated atrial electrogram ablation. Non-PAF initiation and maintenance depend on a critical mass, which allows reentry. The left atrial anterior wall contains a series of substrates that are associated with AF, such as low-voltage zones, Bachmann's bundle, and the LAA, which are important for AF initiation and maintenance. Combining CPVI with left RL, left ASL, and MIL ablation can create a box lesion set on the anterior wall which compartmentalize the left atrial anterior wall into small regions to modify the substrate. We hypothesized that this substrate modification strategy would improve the success rate of non-PAF ablation. However, functional damage to the LAA resulting from the above-mentioned ablation strategy may increase stroke risk. The combined use of AF ablation and LAA occlusion is safe and can reduce stroke risk. Therefore, we examined the safety, feasibility, and efficacy of a new treatment strategy for non-PAF, defined as the CPVI; left ROof linear, Mitral Isthmus linear, and left anterior SEptal linear ablation; and LAA Device occlusion (PROMISED) procedure. Cases were prospectively treated in a 2-arm 1:1 design according to ablation strategy, divided into the Promised group (n = 83) or the PVI combined LAAC group (n =83).

ELIGIBILITY:
Inclusion criteria:

1. Age > 18 years;
2. Persistent AF (AF duration > 7 days);
3. CHA2DS2-VASc score ≥2;
4. Presence of at least one of the following conditions:

   * Unsuitable for long-term standardized anticoagulation therapy;
   * Stroke or embolism still occurred based on long-term standardized anticoagulation therapy;
   * HAS-BLED score ≥3;
   * Unwillingness for long-term anticoagulation therapy;

Exclusion Criteria:

1. Previous atrial fibrillation ablation
2. Transthoracic echocardiography suggests that the anteroposterior diameter of the left atrium is greater than 60 mm;
3. persistent AF that lasts >10 years
4. Scheduled cardiac surgical intervention.
5. Documented left atrial thrombus/ left atrial appendage thrombus or another abnormality that precludes catheter/LAAC introduction
6. Life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-01-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia after a single ablation procedure. | 12 months after the first procedure
  Recurrence rate (percentage) of atrial fibrillation or atrial flutter or atrial tachycardia > 30 seconds after the blanking period of 3-month post ablation, at 1 year after a single ablation procedure. (use of antiarrhythmic medications was not allowed after the blanking period of 3-month)

SECONDARY OUTCOMES:
Recurrence of AF after a single ablation procedure | 12 months after the first procedure
  Recurrence rate (percentage) of AF> 30 seconds after the blanking period of 3 months post ablation, at 1 year after a single ablation procedure. (use of antiarrhythmic medications was not allowed after the blanking period of 3-month)
Recurrence of atrial flutter/atrial tachycardia after a single ablation | 12 months after the first procedure
  Recurrence rate (percentage) of atrial flutter/atrial tachycardia> 30 seconds after the blanking period of 3 months post ablation, at 1 year after a single ablation procedure. (use of antiarrhythmic medications was not allowed after the blanking period of 3-month)
Occurrence of Intra-procedure conversion of persistent AF to sinus rhythm rate and Its Relationship to 1-Year Sinus Rhythm Maintenance Rate | 12 months after the first procedure
  Occurrence of Intra-procedure conversion of persistent AF to sinus rhythm rate (excluding converted to sinus rhythm with cardioversion) and Its Relationship to 1-Year Sinus Rhythm Maintenance Rate
Occurrence of Intra-procedure Conversion from AF to Atrial Flutter or Atrial Tachycardia rate and Its Relationship to 1-Year Sinus Rhythm Maintenance Rate | 12 months after the first procedure
  Occurrence of Intra-procedure Conversion from AF to Atrial Flutter or Atrial Tachycardia rate and Its Relationship to 1-Year Sinus Rhythm Maintenance Rate
Incidence of periprocedural complications | period of Post-operative to hospital discharge
  Incidence of periprocedural complications such as death, pericardial tamponade, stroke, occluder dislodgement, hemorrhage, esophageal injury, complications at access site (hematoma, arteriovenous fistula, pseudoaneurysm)
post-procedure complications | 12 months after the first procedure
  Incidence of post-procedure complications including death, stroke, major bleeding, cardiac tamponade, esophageal injury, and death.
Procedure duration of three-dimensional reconstruction of the left atrial | At the end of the first procedure
  Procedure duration of three-dimensional reconstruction of the left atrial
Procedure duration at ablation | At the end of the first procedure
  Procedure duration at ablation
Procedure duration at LAAC | At the end of the first procedure
  Procedure duration at LAAC
Incidence of events including device-related thrombus and peri-device leak at 3 months post-procedure | 3 months after the first procedure
  Incidence of events including device-related thrombus and peri-device leak at 3 months post-procedure
Anticoagulant discontinuation rate at 6 months post-procedure | 6 months after the first procedure
  Anticoagulant discontinuation rate at 6 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yue-chun Li, MD, Principal Investigator — Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University
Locations (1):
- Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China